CLINICAL TRIAL: NCT05471141
Title: Preventing and Managing Cognitive Impairment
Acronym: CognitnECHO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty obtaining IRB approval from all sites with challenges in recruitment. No participants enrolled. So, we revised the study. Now it does not meet the NIH or FDA's definition of clinical trials. We request to close this registration.
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1931012
Record Dates: First submitted 2022-06-30; First posted 2022-07-22 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Knowledge Translation; Cognitive Impairment
Keywords: primary health care; cognitive impairment; translational science; translational research; general practitioners; Minority Health
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Group 1 will receive the intervention Cognition ECHO during Phase 1 and Group 2 will serve as the control. About one month after Group 1 has completed the attendance of all five sessions of Cognition ECHO, Group 2 will start receiving the intervention Cognition ECHO and Group 1 will wait for the follow-up till Week 41 of the study in November 2023.
Who Masked: Participant
Masking Description: All participants will be informed that they will receive intervention but one group starts first and the other group will start with a 4-month delay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): To receive intervention during the phase 1 and will receive nothing during the phase 2, will complete the measure at the end of phase 2 as the follow-up
  Interventions: Other: Cognition ECHO
- Group 2 (No Intervention): To serve as the control during phase 1 and receive intervention during the phase 2

INTERVENTIONS:
Other: Cognition ECHO — Cognition ECHO is the intervention designed to be used by the study participants who are primary care practitioners. No involvement of patients in this study. The panel will consist of the CI and Co-PIs of this study, a neurologist as a co-moderator, a medical specialist who is the expert on the subject, an occupational therapist, a psychologist, and a speech and language pathologist with experience and expertise in CI. A patient with CI and a caregiver, family member, or community representative who is not a healthcare professional will join the panel because CI is frequently observed with lived experience of family members and loved ones, as two non-clinician panelists. The five topics with the integration of related diagnoses for Cognition ECHO are listed in Table 4. The time allocated for the didactic will be 15-20 minutes and the de-identified case discussion will be 40 - 45 minutes.
  Other Names: Tele-mentoring with (1) a didactic presentation and (2) de-identified discussion by a panel with experts, a patient, and a family member.
  Arms: Group 1

SUMMARY:
This randomized controlled trial (RCT) is used to address the knowledge translation of primary care practitioners (PCPs) for the early identification of cognitive impairment. Cognitive impairment is experienced by people with many different underlying health problems, e.g., diabetes, cardiovascular problems, COVID-19, neurodegenerative diseases, and mental health problems. Older adults are more likely to have cognitive decline which may develop into Alzheimer's disease or dementia but 40% of dementia can be prevented by managing the risks. Cognitive impairment can demand vast societal resources, the burden is reported to be more among Hispanics and blacks. By 2029, all baby boomers will be over 65, comprising at least 20% of the U.S. population. So, it is critical for PCPs to effectively identify, prevent, and manage the hidden signs of cognitive impairment. People with early signs of cognitive impairment will have opportunities to benefit from suitable cognitive remediation to reverse it or prevent rapid progression. It is critically important for people who are socioeconomically disadvantaged, those who are black, indigenous, and people of color (BIPoC). These people are often served by safety-net hospitals, such as clinics of the Los Angeles County (LAC) Department of Health Services and the federally qualified health centers at the Community Clinics Association of LAC. Many PCPs in these clinics are often BIPoC. The intervention used in this RCT is called "Cognition ECHO" based on the proven model of ECHO (Extension of Healthcare Outcomes) for knowledge dissemination and translation. Cognition ECHO is a virtual activity incorporating a short didactic presentation and de-identified case discussion to solve real-world patient care challenges and ease direct knowledge translation. PCPs in the LAC will be randomized into Groups 1 and 2. Group 1 will attend the five Cognition ECHO for four months, Group 2 will be the control. Group 2 will attend Cognition ECHO starting on July 25, 2023, five times till November 7, 2023, when Group 1 is the follow-up. Most sessions are scheduled on the fourth Tuesday of the month with the addition of June 6 and November 7, 2023. Focusing on cognitive impairment and targeting PCPs at the LAC, the goal of this study is to evaluate if Cognition ECHO can improve PCPs' capacity to detect early cognitive impairment and manage it. It will result in opportunities to mitigate the risk factors of early cognitive impairment, especially for minority patients in LAC, and conduct efficacy studies in the future to address cognitive impairment focusing on BIPoC.

ELIGIBILITY:
Inclusion Criteria:

1. Primary care practitioner (i.e. physician, NP or PA) at least 21-year-old.
2. Spending at least 40% of the work hours in patient care with adult patients currently.
3. Self-identifying being comfortable to attend virtual learning sessions using their own smartphones, laptops/desktop computers, or mobile devices in their work setting.
4. Willingness to send in a total of four electronic copies (in WORD) of de-identified clinic notes written documenting the initial encounters of patients with poorly controlled type 2 diabetes (A1c >= 8%) or any patients with early signs of neurodegenerative diseases, Alzheimer's diseases or other conditions that may affect the cognition.

Exclusion Criteria:

* Do not work at least 40% of the week for care provision in primary care
* Do not work in the outpatient clinics of the Los Angeles County (LAC) Department of Health Services (DHS) and member clinics of the Community Clinics of the Los Angeles County (CCALAC) with the federally qualified health centers (FQHCs).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-13 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Estimated adherence1 | The 2nd day of Week 9 to the end of Week 9 for Group 1. The 2nd day of Week 26 to the end of Week 26 for Group 2.
  The ETAC (Empowered-To-Act Consistently) scale is used to measure the estimated adherence. The categories are to guide learners' reflection on their future actions, not measuring change. Four ETAC questions are designed for the four cognition management tasks to be included in a post-session evaluation of a Cognition ECHO session. Using the ETAC scale, the reasons and concerns of the option selected can be explored qualitatively. The ETAC scale has six levels:
  A) I will not do it; because: _. B) I will think about it, because: _. C) I will think about ways to help me start doing it, specific areas: _ . D) I'll start doing it from now on, areas to start: _. E) I've done some but can still do more, areas to do more: _. F) I am doing it as much as I can. No new actions are needed; sharing your successful experience: _.
  The percentages of those picked options C, D, and E will be used in this study as estimated adherence for each session of the Cognition ECHO.
Estimated adherence2 | The 2nd day of Week 13 to the end of Week 13 for Group 1; the 2nd day of Week 30 to the end of Week 30 for Group 2.
  The ETAC (Empowered-To-Act Consistently) scale is used to measure the estimated adherence. The categories are to guide learners' reflection on their future actions, not measuring change. Four ETAC questions are designed for the four cognition management tasks to be included in a post-session evaluation of a Cognition ECHO session. Using the ETAC scale, the reasons and concerns of the option selected can be explored qualitatively. The ETAC scale has six levels:
  A) I will not do it; because: _. B) I will think about it, because: _. C) I will think about ways to help me start doing it, specific areas: _ . D) I'll start doing it from now on, areas to start: _. E) I've done some but can still do more, areas to do more: _. F) I am doing it as much as I can. No new actions are needed; sharing your successful experience: _.
  The percentages of those picked options C, D, and E will be used in this study as estimated adherence for each session of the Cognition ECHO
Estimated adherence3 | The 2nd day of Week 17 to the end of Week 17 for Group 1; the 2nd day of Week 35 to the end of Week 35 for Group 2.
  The ETAC (Empowered-To-Act Consistently) scale is used to measure the estimated adherence. The categories are to guide learners' reflection on their future actions, not measuring change. Four ETAC questions are designed for the four cognition management tasks to be included in a post-session evaluation of a Cognition ECHO session. Using the ETAC scale, the reasons and concerns of the option selected can be explored qualitatively. The ETAC scale has six levels:
  A) I will not do it; because: _. B) I will think about it, because: _. C) I will think about ways to help me start doing it, specific areas: _ . D) I'll start doing it from now on, areas to start: _. E) I've done some but can still do more, areas to do more: _. F) I am doing it as much as I can. No new actions are needed; sharing your successful experience: _.
  The percentages of those picked options C, D, and E will be used in this study as estimated adherence for each session of the Cognition ECHO
Estimated adherence4 | The 2nd day of Week 19 to the end of Week 19 for Group 1; the 2nd day of Week 39 to the end of Week 39 for Group 2.
  The ETAC (Empowered-To-Act Consistently) scale is used to measure the estimated adherence. The categories are to guide learners' reflection on their future actions, not measuring change. Four ETAC questions are designed for the four cognition management tasks to be included in a post-session evaluation of a Cognition ECHO session. Using the ETAC scale, the reasons and concerns of the option selected can be explored qualitatively. The ETAC scale has six levels:
  A) I will not do it; because: _. B) I will think about it, because: _. C) I will think about ways to help me start doing it, specific areas: _ . D) I'll start doing it from now on, areas to start: _. E) I've done some but can still do more, areas to do more: _. F) I am doing it as much as I can. No new actions are needed; sharing your successful experience: _.
  The percentages of those picked options C, D, and E will be used in this study as estimated adherence for each session of the Cognition ECHO
Estimated adherence5 | The 2nd day of Week 22 to the end of Week 22 for Group 1; the 2nd day of Week 41 to the end of Week 41 for Group 2.
  The ETAC (Empowered-To-Act Consistently) scale is used to measure the estimated adherence. The categories are to guide learners' reflection on their future actions, not measuring change. Four ETAC questions are designed for the four cognition management tasks to be included in a post-session evaluation of a Cognition ECHO session. Using the ETAC scale, the reasons and concerns of the option selected can be explored qualitatively. The ETAC scale has six levels:
  A) I will not do it; because: _. B) I will think about it, because: _. C) I will think about ways to help me start doing it, specific areas: _ . D) I'll start doing it from now on, areas to start: _. E) I've done some but can still do more, areas to do more: _. F) I am doing it as much as I can. No new actions are needed; sharing your successful experience: _.
  The percentages of those picked options C, D, and E will be used in this study as estimated adherence for each session of the Cognition ECHO
The "System Usability Scale of Cognition Management Tasks" (SUS CMTs) - 1 | Week 4 to Week 8, Baseline.
  The System Usability Scales of Cognitive Management Tasks (SUS CMTs) are adapted from the standardized measure, System Usability Scale. Each scale has ten items and a five-point scale ranging from "strongly disagree" to "strongly agree." The final score ranges from 0 to 100. A high score indicates high usability. The SUS CMTs are used to measure the perceived usability of the cognitive management tasks.
The "System Usability Scale of Cognition Management Tasks" (SUS CMTs) - 2 | The 2nd day of Week 22 to the end of Week 25
  The System Usability Scales of Cognitive Management Tasks (SUS CMTs) are adapted from the standardized measure, System Usability Scale. Each scale has ten items and a five-point scale ranging from "strongly disagree" to "strongly agree." The final score ranges from 0 to 100. A high score indicates high usability. The SUS CMTs are used to measure the perceived usability of the cognitive management tasks.
The "System Usability Scale of Cognition Management Tasks" (SUS CMTs) - 3 | The 2nd day of Week 41 to the end of Week 44
  The System Usability Scales of Cognitive Management Tasks (SUS CMTs) are adapted from the standardized measure, System Usability Scale. Each scale has ten items and a five-point scale ranging from "strongly disagree" to "strongly agree." The final score ranges from 0 to 100. A high score indicates high usability. The SUS CMTs are used to measure the perceived usability of the cognitive management tasks.
The "Self-Efficacy of Cognition Management Tasks" - 1 | The 2nd day of Week 22 to the end of Week 25
  The Self-Efficacy of Cognition Management Tasks (CMTs) is a survey adapted from a self-efficacy scale for primary care practitioners to evaluate their self-efficacy in diabetes care provision (Bouchonville et al., 2018). The Self-Efficacy of CMTs measures the capacity of PCPs to do these cognition management tasks. It is a survey with ten items using a seven-point scale ranging from "none, no skills" to "expert, teaching others." The final score ranges from 10 to 70 with a high score reflecting better self-efficacy. The items reflect the knowledge and skills most relevant to detecting and managing cognitive impairment by primary care practitioners. With the adjustment to address response shift bias, the retrospective pre-intervention status will be compared together.
The "Self-Efficacy of Cognition Management Tasks" - 2 | The 2nd day of Week 41 to the end of Week 44
  The Self-Efficacy of Cognition Management Tasks (CMTs) is a survey adapted from a self-efficacy scale for primary care practitioners to evaluate their self-efficacy in diabetes care provision (Bouchonville et al., 2018). The Self-Efficacy of CMTs measures the capacity of PCPs to do these cognition management tasks. It is a survey with ten items using a seven-point scale ranging from "none, no skills" to "expert, teaching others." The final score ranges from 10 to 70 with a high score reflecting better self-efficacy. The items reflect the knowledge and skills most relevant to detecting and managing cognitive impairment by primary care practitioners. With the adjustment to address response shift bias, the retrospective pre-intervention status will be compared together.

SECONDARY OUTCOMES:
Changes seen through the evidence of cognition management tasks in clinical encounter notes | the baseline two -identified clinic encounter notes: Baseline (30 days). Post-intervention (30 days).
  Evidence of CMTs in clinical encounter notes will be explored using artificial intelligence, natural language processing (NLP) method. It is a machine learning process for the project team to develop the list of words and phrases related to CMTs to be included in machine learning and to perform the search, to extract, organize, and aggregate evidence of CMTs embedded in the de-identified clinic encounter notes.

CONTACTS AND LOCATIONS:
Overall Officials: Shan-Pin C Fanchiang, Ph.D., Principal Investigator — Charles Drew University of Medicine and Science

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and the Clinical Study Report.
Supporting Information: Study Protocol, CSR
Time Frame: Both items will be available to share from January 5, 2025, to June 30, 2025.
Access Criteria: By sending an email request to the PI, shanpinfanchiang@cdrewu.edu.